CLINICAL TRIAL: NCT00686712
Title: The Utility of Insulin Glargine (Lantus) Compared to NPH in Ethnic Minority Type 2 Diabetic Subjects Starting Insulin Therapy
Brief Title: Insulin Glargine at Bedtime or in AM Versus NPH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 03-02-524; U54RR014616 (NIH)
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2010-10-07 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Glargine; Type 2 diabetes; Basal insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Drugs, Generic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 - Insulin glargine QHS (Experimental): Insulin glargine injected subcutaneously once daily at bedtime
  Interventions: Drug: 1- Insulin glargine QHS
- 2 - Insulin glargine QAM (Experimental): Insulin glargine injected subcutaneously once daily in the morning
  Interventions: Drug: 2 - Insulin glargine QAM
- 3 - NPH Insulin QHS (Active Comparator): NPH insulin injected subcutaneously once daily at bedtime
  Interventions: Drug: 3 - NPH insulin QHS

INTERVENTIONS:
Drug: 1- Insulin glargine QHS — Insulin glargine at bedtime (dose titrated to maintain 50% of fasting glucose readings <120 mg/dL)
  Other Names: Trade name: Lantus
  Arms: 1 - Insulin glargine QHS
Drug: 2 - Insulin glargine QAM — Insulin glargine in AM (dose titrated to maintain 50% of pre-supper glucose readings <120 mg/dL)
  Other Names: Trade name: Lantus
  Arms: 2 - Insulin glargine QAM
Drug: 3 - NPH insulin QHS — NPH insulin at bedtime (dose titrated to maintain 50% of fasting glucoses <120 mg/dL)
  Other Names: (Generic)
  Arms: 3 - NPH Insulin QHS

SUMMARY:
To compare the efficacy and safety of once-nightly insulin glargine versus a single morning injection of glargine or once-nightly NPH insulin in ethnic minority type 2 diabetic patients inadequately controlled on combination oral agents.

DETAILED DESCRIPTION:
Insulin glargine has a longer action than compared to NPH insulin, but whether this results in improved control when used as a once-nightly or morning basal insulin injection in type 2 diabetic patients who are inadequately controlled on combination oral agents has been controversial. Inner city ethnic minority patients with diabetes are a particularly challenging population of diabetic patients to treat. This study investigates whether insulin glargine may be a more effective or safer first-line basal insulin than NPH in this population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-75
* Type 2 diabetes diagnosed for at least 1 year
* Treatment with stable doses of oral agents (alone or in combination) for at least 2 months
* Inadequate glycemic control (hemoglobin A1c ≥ 7.5%) on maximum-tolerated doses of a sulfonylurea, metformin and a thiazolidinedione
* No past history of chronic insulin use (other than treatment of gestational diabetes or hospitalizations of less than 1 week in duration)
* Hemoglobin A1c between 7.5% and 12%
* Body mass index (BMI) between 20 and 40 kg/m2

Exclusion Criteria:

* Current or previous chronic use of insulin (other than for treatment of gestational diabetes)
* History of confirmed (or clinical suspicion of) type 1 diabetes
* Female subjects of childbearing potential who are sexually active and not using a reliable form of contraception
* Current pregnancy or lactation.
* Subjects for whom insulin therapy is contraindicated or for whom, in the opinion of the investigator, therapy with insulin is not indicated
* Subjects with advanced proliferative diabetic retinopathy
* Subjects who work night shifts or who are unable to stay on a consistent daily meal schedule
* History of any clinically significant renal, hepatic, cardiovascular, neurological, endocrinological or other major systemic disease that, in the opinion of the investigator, may make implementation of the protocol or interpretation of the data difficult.
* Subjects who will likely require or initiate therapy with drugs which may interfere with glucose metabolism during the course of the study
* Subjects who are in another investigational study or have received another investigational medication within 30 days of study entry
* Subjects who are unable or unwilling to comply with all components of the study protocol, including contacting the investigators at specified times and attending all scheduled follow-up visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2003-02; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Hsia, MD, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles Drew University of Medicine and Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Semlitsch T, Engler J, Siebenhofer A, Jeitler K, Berghold A, Horvath K. (Ultra-)long-acting insulin analogues versus NPH insulin (human isophane insulin) for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Nov 9;11(11):CD005613. doi: 10.1002/14651858.CD005613.pub4. PMID 33166419
- [Derived] Hsia SH. Insulin glargine compared to NPH among insulin-naive, U.S. inner city, ethnic minority type 2 diabetic patients. Diabetes Res Clin Pract. 2011 Mar;91(3):293-9. doi: 10.1016/j.diabres.2010.11.028. Epub 2010 Dec 13. PMID 21146881

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred from Sep 2002 to Feb 2009. Subjects recruited from a diabetes specialty referral clinic, as well as from primary care clinics and through advertising in the South Los Angeles area.
Pre-assignment Details: Baseline run-in period to document baseline control and reinforce dietary/lifestyle principles.
  23 subjects not randomized due to protocol violations, loss to follow-up, lack of need for insulin, or voluntarily.
Groups:
- Insulin Glargine at Bedtime: Bedtime insulin glargine titrated to morning fasting glucose readings
- Insulin Glargine in AM: Morning insulin glargine titrated to pre-supper glucose readings
- NPH Insulin: Bedtime NPH insulin titrated to morning fasting glucose readings
Period: Overall Study
Arm/Group | Insulin Glargine at Bedtime | Insulin Glargine in AM | NPH Insulin
Started | 30 | 25 | 30
Completed | 20 | 14 | 17
Not Completed | 10 | 11 | 13
Not completed — Protocol Violation | 8 | 8 | 10
Not completed — Lost to Follow-up | 1 | 2 | 3
Not completed — Adverse Event | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin Glargine at Bedtime | Insulin Glargine in AM | NPH Insulin | Total
Number analyzed (Participants) | 30 | 25 | 30 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (11.2) | 53.0 (8.6) | 53.2 (7.7) | 52.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 13 | 21 | 49
  Male | 15 | 12 | 9 | 36
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 24 | 21 | 25 | 70
  Not Hispanic or Latino | 6 | 4 | 5 | 15
Hemoglobin A1c [Mean (Standard Deviation); unit: Percent] | 9.2 (1.3) | 9.6 (1.2) | 9.3 (1.6) | 9.3 (1.4)
Diabetes Duration [Mean (Standard Deviation); unit: Years] | 9.0 (5.9) | 9.5 (5.2) | 7.8 (4.2) | 8.7 (5.1)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.6 (5.0) | 31.1 (5.2) | 32.1 (6.0) | 31.6 (5.4)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c Change From Baseline
Time Frame: Baseline to 6 months
Population: ITT (LOCF)
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Insulin Glargine at Bedtime | Insulin Glargine in AM | NPH Insulin
Number analyzed (Participants) | 30 | 25 | 30
Percent | -1.3 (1.2) | -1.9 (1.4) | -1.4 (1.7)

2. Secondary Outcome: Frequency of Glucose Readings < 130 mg/dL
Description: Frequency of glucose readings below the recommended pre-meal glucose target of 130 mg/dL
Time Frame: 6 months
Population: Enrolled subjects
Measure: Mean (Standard Deviation); unit: percentage of readings
Groups:
- 1 - Insulin Glargine QHS: Insulin glargine injected subcutaneously once daily at bedtime
  Insulin glargine injected subcutaneously once daily at bedtime: Insulin glargine at bedtime (dose titrated to maintain 50% of fasting glucose readings <120 mg/dL)
- 2 - Insulin Glargine QAM: Insulin glargine injected subcutaneously once daily in the morning
  Insulin glargine injected subcutaneously once daily in the morning: Insulin glargine in AM (dose titrated to maintain 50% of pre-supper glucose readings <120 mg/dL)
- 3 - NPH Insulin QHS: NPH insulin injected subcutaneously once daily at bedtime
  NPH insulin injected subcutaneously once daily at bedtime: NPH insulin at bedtime (dose titrated to maintain 50% of fasting glucoses <120 mg/dL)
Arm/Group | 1 - Insulin Glargine QHS | 2 - Insulin Glargine QAM | 3 - NPH Insulin QHS
Number analyzed (Participants) | 30 | 25 | 30
percentage of readings | 61.7 (22.8) | 73.0 (25.1) | 72.6 (22.7)

3. Secondary Outcome: Frequency of Total Hypoglycemic Reactions
Description: Frequency of hypoglycemic reactions without regard to time of occurrence
Time Frame: 6 months
Population: Enrolled subjects
Measure: Mean (Standard Deviation); unit: Hypoglycemic events per patient
Arm/Group | 1 - Insulin Glargine QHS | 2 - Insulin Glargine QAM | 3 - NPH Insulin QHS
Number analyzed (Participants) | 30 | 25 | 30
Hypoglycemic events per patient | 6.7 (9.6) | 9.6 (6.6) | 8.2 (8.7)

4. Secondary Outcome: Frequency of Severe Hypoglycemic Reactions
Description: Frequency of severe hypoglycemic reactions, defined as those requiring the assistance of another person
Time Frame: 6 months
Population: Enrolled subjects
Measure: Number; unit: Severe hypoglycemic events
Arm/Group | 1 - Insulin Glargine QHS | 2 - Insulin Glargine QAM | 3 - NPH Insulin QHS
Number analyzed (Participants) | 30 | 25 | 30
Severe hypoglycemic events | 0 | 0 | 0

5. Secondary Outcome: Body Mass Index Change From Baseline
Description: Change in body mass index from baseline BMI measurement
Time Frame: 6 months
Population: Enrolled subjects
Measure: Mean (Standard Deviation); unit: kg per square meter
Arm/Group | 1 - Insulin Glargine QHS | 2 - Insulin Glargine QAM | 3 - NPH Insulin QHS
Number analyzed (Participants) | 30 | 25 | 30
kg per square meter | 0.7 (1.6) | 1.1 (1.4) | 0.0 (1.5)

6. Secondary Outcome: Total Daily Insulin Dose
Description: Total daily number of units of insulin used
Time Frame: 6 months
Population: Enrolled subjects
Measure: Mean (Standard Deviation); unit: Units of insulin per day
Arm/Group | 1 - Insulin Glargine QHS | 2 - Insulin Glargine QAM | 3 - NPH Insulin QHS
Number analyzed (Participants) | 30 | 25 | 30
Units of insulin per day | 17.7 (10.1) | 17.9 (14.4) | 14.6 (13.4)

7. Secondary Outcome: Any Adverse Event Other Than Hypoglycemia
Description: Any reported adverse event that is not hypoglycemia
Time Frame: 6 months
Population: Enrolled subjects
Measure: Number; unit: Events
Arm/Group | 1 - Insulin Glargine QHS | 2 - Insulin Glargine QAM | 3 - NPH Insulin QHS
Number analyzed (Participants) | 30 | 25 | 30
Events | 1 | 2 | 1

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Insulin Glargine at Bedtime | Insulin Glargine in AM | NPH Insulin
Serious Adverse Events (participants affected / at risk) | 0/30 | 1/25 | 0/30
Other Adverse Events (participants affected / at risk) | 23/30 | 24/25 | 23/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine at Bedtime (N=30) | Insulin Glargine in AM (N=25) | NPH Insulin (N=30)
Foot Infection (Hospitalization) (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin Glargine at Bedtime (N=30) | Insulin Glargine in AM (N=25) | NPH Insulin (N=30)
Symptomatic Hypoglycemia (Endocrine disorders) | 23 (200) | 24 (239) | 23 (247) — Classic symptoms of hypoglycemia, relieved by carbohydrate ingestion, with or without a corroborating self-monitored glucose reading
Asymptomatic Retinal Hemorrhage (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to smaller than anticipated enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes